CLINICAL TRIAL: NCT06372431
Title: Multicenter, Non-interventional Observational Prospective Study With Retrospective Analysis to Describe the Rate of CKD Diagnosis, in Patients With Arterial Hypertension and CKD Markers
Brief Title: PRospectIve ObseRvatIonal mulTicenter Study of Patients With Arterial hYpertension and CKD in the Population of Russia
Acronym: PRIORITY-CKD
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1843R00360
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Arterial Hypertension, Chronic Kidney Disease
Keywords: arterial hypertension, chronic kidney disease, CKD, AH
MeSH Terms: conditions — Hypertension; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a multi-centre, non-interventional, observational, prospective study with retrospective analysis. The main purpose of the study is to describe the rate of CKD diagnosis in patients with AH and CKD markers. This study will include 10 000 adult outpatients with arterial hypertension, who have one or more Chronic Kidney Disease laboratory markers (without recorded CKD diagnosis prior to enrolment) and have no diabetes mellitus or symptomatic chronic heart failure, who are monitored and treated by cardiologists or internal medicine specialists in approximately 50 outpatient sites in about 20 regions in Russia.

This observational study does not provide for any diagnostic and therapeutic procedures other than those used in routine practice.

DETAILED DESCRIPTION:
Timely chronic kidney disease (CKD) detection is important for slowing or preventing of kidney function deterioration, reducing cardiovascular complications and mortality. Unfortunately, early-stage CKD is primarily asymptomatic, and due to lack of symptoms CKD is often diagnosed only in advanced stages.

There are limited epidemiological data of the overall CKD prevalence in Russia. In Russia there is Federal diabetes registry that includes data of diabetes kidney disease among others, so the population of patients with diabetes mellitus (DM) and CKD is more studied. Besides the diabetes, AH is also considered one of the major etiological factors for CKD development and progression, but the population of patients with AH and CKD is less studied. Available studies that assess renal function in patients with AH are cross-sectional with one-time assessment of kidney function. The diagnosis of CKD should be established, if CKD markers are observed over 3 or more months, so it is required to assess the markers of kidney function and/or kidney damage overtime to confirm chronic condition.

There is a need to conduct a large observational study in patients with AH and CKD markers to describe the rate of CKD diagnosis in this patient population. Recorded diagnosis of CKD is an important first step to reduce the risk of disease progression and minimize adverse clinical outcomes.

The current study will enroll patients with AH and without previously diagnosed DM and symptomatic heart failure that will allow focusing on evaluating the prevalence of newly diagnosed CKD in patients with hypertension.

This study is a multi-center, non-interventional, observational, prospective study with retrospective analysis.

Planned study population for prospective analysis consists of 10 000 adult outpatients with AH and one or more CKD markers, without recorded CKD diagnosis prior to enrolment, and without recorded diagnosis of DM or symptomatic chronic heart failure (CHF). Planned number of study sites is approximately 50 outpatient sites in about 20 regions of Russia.

Retrospective part includes retrospective review by the physician of paper or electronic medical records of patients with recorded diagnosis of AH for the presence of laboratory CKD markers, measured within the period of ≤12 months prior to inclusion into the study. Patients with one or more CKD markers recorded in their medical records (without recorded CKD diagnosis) can be included in the prospective part of the study.

Demographic and clinical characteristics, including medical history, CKD markers, will be collected retrospectively from all enrolled patients.

In case of enough retrospective data for the period of ≤12 months prior to inclusion to confirm CKD diagnosis according to the current clinical guidelines (two consecutive evaluations of CKD marker(s) with the interval between two measurements not less than 3 months), the CKD diagnosis can be confirmed and recorded. Otherwise, the laboratory testing will be performed to confirm or exclude the CKD diagnosis.

Overall expected duration of the study (from the first patient inclusion to the last patient last visit) is 18 months, or until 10 000 eligible patients are included to the study and data on these patients are collected, whichever occurs first.

This non-interventional study does not imply any intervention into a routine clinical practice, and does not provide for any diagnostic and therapeutic procedures other than those used in routine practice.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants aged 18 years or older at the time of signing the ICF;
2. Signed and dated written informed consent in accordance with ICH GCP and local law prior to inclusion in the study;
3. Diagnosis of AH (essential hypertension) previously established in accordance with current Russian "Clinical guidelines on arterial hypertension in adults", i.e. office systolic blood pressure (SBP) ≥140 mmHg and/or diastolic blood pressure (DBP) ≥90 mmHg, measured on two different visits;
4. Laboratory markers of CKD (eGFR < 60 ml/min/1,73 m2 and/or albuminuria/proteinuria*), measured for the period of ≤12 months prior to enrolment. *any of the following: urine ACR (albumin/creatinine ratio) ≥ 30 mg/g (3 mg/mmol), urine PCR (protein/creatinine ratio) ≥150 mg/g (15 mg/mmol), 24-h albuminuria ≥30 mg/day or 24-h proteinuria ≥ 0.15 g/day.
5. No CKD diagnosis recorded in a patient's medical documents prior to enrollment

Exclusion Criteria:

1. The diagnosis of symptomatic chronic heart failure (CHF) II-IV functional class according to the NYHA classification ever recorded in a patient's medical documents;
2. The diagnosis of diabetes mellitus (DM type 1 or DM type 2) recorded in a patient's medical documents;
3. The diagnosis of AH of secondary origin;
4. Participation in any randomized controlled trial within 3 months before the inclusion in this study or during the participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 10 000 adult outpatients with AH, who have one or more CKD laboratory markers (without recorded CKD diagnosis prior to enrolment), and have no DM or CHF, who are monitored and treated by cardiologists or internal medicine specialists
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
To describe the rate of CKD diagnosis in patients with AH and CKD markers. | up to 18 months
  1. Proportion of patients with AH and CKD markers and recorded CKD diagnosis based on retrospective data on Visit 1 ; See Note #1 below.
  2. Proportion of patients with AH and CKD markers with confirmed and recorded CKD diagnosis during Visit 2.
  3. Proportion of patients with AH and CKD markers to whom CKD diagnosis was not confirmed during Visit 2;
  4. Total proportion of patients with confirmed CKD diagnosis in the study, i.e. during Visit 1 or Visit 2.
  Note #1: During Visit 1 (inclusion in the study) the demographic and clinical characteristics, including medical history, CKD markers, will be collected retrospectively from all enrolled patients. In case of enough retrospective data for the period of ≤12 months prior to inclusion to confirm CKD diagnosis according to the current clinical guidelines (two consecutive evaluations of CKD marker(s) with the interval between two measurements not less than 3 months), the CKD diagnosis can be confirmed and recorded during Visit 1.

SECONDARY OUTCOMES:
To describe demographic and clinical characteristics of patients with AH and CKD markers | 18 months
  1. Mean age (years) at the Visit 1, and proportion of patients by age groups;
  2. Proportion of men and women;
  3. Proportion of patients with negative lifestyle factors;
  4. Mean body mass index and proportion of patients with overweight and obesity;
  5. Mean waist circumference (cm) in men and women;
  6. Mean and median duration of AH;
  7. Proportion of patients with various AH stage (I, II, III) and CV risk category (low, moderate, high, very high);
  8. Mean BP (systolic and diastolic) on Visit 1 and Visit 2;
  9. Proportion of patients with uncontrolled AH based on any evaluation during the study (endpoint is assessed in patients who were taking any AH medication); etc
  10. Proportion of patients with resistant AH based on any evaluation during the study
  11. Proportion of patients with CV comorbidities and complications of AH.
To describe clinical characteristics of patients with AH and diagnosed CKD during this study (on Visit 1 or Visit 2) and profile of routine therapy before and after CKD diagnosis | 18 months
  12. Mean values of laboratory parameters; 13. Proportion of patients with presence of abnormalities in urinalysis; 14. Proportion of patients with laboratory investigations abnormalities; 15. Proportion of patients with other concomitant diseases (kidney and urinary tract, systemic connective tissue and oncological); 16. Mean eGFR, ml/min/1.73 m2; 17. Proportion of patients with eGFR ≤59 ml/min/1,73 m2; 18. Proportion of patients with each eGFR category; 19. Proportion of patients with albuminuria categories; 20. Proportion of patients with proteinuria categories; 21. Proportion of patients with each category of risk for prognosis of CKD according to KDIGO; 22. Proportion of patients with ECG signs of left ventricular hypertrophy; 23. Proportion of patients with prestage of CHF; 24. Proportion of patients with signs of changes after ultrasound of the kidney etc.

CONTACTS AND LOCATIONS:
Locations (30):
- Russia (30):
  - Research Site, Aramil
  - Research Site, Chelyabinsk
  - Research Site, Irkutsk
  - Research Site, Kaluga
  - Research Site, Kazan'
  - Research Site, Kemerovo
  - Research Site, Krasnodar
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Odintsovo
  - Research Site, Omsk
  - Research Site, Penza
  - Research Site, Perm
  - Research Site, Reutov
  - Research Site, Rostov-on-Don
  - Research Site, Ryazan
  - Research Site, Saint Petersburg
  - Research Site, Samara
  - Research Site, Stavropol
  - Research Site, Tomsk
  - Research Site, Tula
  - Research Site, Ufa
  - Research Site, Ulan-Ude
  - Research Site, Volgograd
  - Research Site, Vologda
  - Research Site, Voronezh
  - Research Site, Yaroslavl
  - Research Site, Yekaterinburg